CLINICAL TRIAL: NCT00002785
Title: Treatment of Newly Diagnosed Acute Lymphoblastic Leukemia in Infants Less Than 1 Year of Age.
Brief Title: Combination Chemotherapy, Bone Marrow Transplantation, and Radiation Therapy in Treating Infants With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1953; CCG-1953 (Other: Children's Cancer Group); CDR0000064841 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Filgrastim; Asparaginase; Cyclophosphamide; Cyclosporine; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Leucovorin; Mercaptopurine; Mesna; Methotrexate; Methylprednisolone; pegaspargase; Prednisone; Hydrocortisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: asparaginase
Drug: cyclophosphamide
Drug: cyclosporine
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: leucovorin calcium
Drug: mercaptopurine
Drug: mesna
Drug: methotrexate
Drug: methylprednisolone
Drug: pegaspargase
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Procedure: allogeneic bone marrow transplantation
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Bone marrow transplantation may allow the doctor to give higher doses of chemotherapy and kill more cancer cells. Radiation therapy uses high-energy x-rays to damage cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, bone marrow transplantation, and radiation therapy in treating infants with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the feasibility and outcome of intensified induction/consolidation followed by intensified re-induction/re-intensification in infants less than 1 year of age with newly diagnosed acute lymphocytic leukemia (ALL). II. Evaluate the feasibility and outcome of bone marrow transplantation using family or unrelated donors in infants with the 11q23 abnormality. III. Evaluate neuropsychologic outcome upon completion of protocol therapy in patients who have reached the ages of 3 and 7 years, with special attention to the outcome in infants who received total-body irradiation. IV. Study the biology of infant ALL in samples of leukemic blood and bone marrow. V. Study the possible associations among patient- and disease-specific factors and family sociodemographic characteristics that mediate treatment outcome.

OUTLINE: Upon completion of Induction/Intensification and Re-Induction therapy, patients with the 11q23 abnormality and with a matched or one-antigen mismatched related or unrelated donor proceed immediately to Transplantation; all others proceed to Re-Intensification, Consolidation, Intensified Maintenance, and Routine Maintenance. The following acronyms are used: AlBM Allogeneic Bone Marrow ARA-C Cytarabine, NSC-63878 ASP Asparaginase, NSC-109229 CF Leucovorin calcium, NSC-3590 CTX Cyclophosphamide, NSC-26271 CYSP Cyclosporine, NSC-290193 DM Dexamethasone, NSC-34521 DNR Daunorubicin, NSC-82151 G-CSF Granulocyte-Colony Stimulating Factor (Amgen), NSC-614629 HC Hydrocortisone, NSC-10483 MePRDL Methylprednisolone, NSC-19987 Mesna Mercaptoethane sulfonate, NSC-113891 MP Mercaptopurine, NSC-755 MTX Methotrexate, NSC-740 PEG-ASP Pegaspargase, NSC-644954 PRED Prednisone, NSC-10023 TBI Total-Body Irradiation TIT Triple Intrathecal Therapy (IT ARA-C/IT HC/IT MTX) VCR Vincristine, NSC-67574 VH Very High Dose VP-16 Etoposide, NSC-141540 INDUCTION/INTENSIFICATION: 5-Drug Combination Systemic Chemotherapy followed by 3-Drug Combination Systemic Chemotherapy plus 3-Drug Combination Intrathecal Chemotherapy. DM/VCR/DNR/CTX/Mesna/ASP; followed by MTX/CF/VP-16/CTX/Mesna; plus TIT. RE-INDUCTION: 5-Drug Combination Systemic Chemotherapy plus 3-Drug Combination Intrathecal Chemotherapy. DNR/VCR/CTX/Mesna/ASP/DM; plus TIT. RE-INTENSIFICATION: 2-Drug Combination Systemic Chemotherapy plus Single-Agent Intrathecal Chemotherapy followed by 2-Drug Combination Systemic Chemotherapy. VCR/VH MTX/CF; plus IT ARA-C; followed by VP-16/CTX/Mesna. CONSOLIDATION: 2-Drug Combination Systemic Chemotherapy followed by 2-Drug Combination Systemic Chemotherapy plus Single-Agent Intrathecal Chemotherapy. ARA-C/ASP; followed by VH MTX/CF/VCR; plus IT ARA-C. INTENSIFIED MAINTENANCE: 4-Drug Combination Systemic Chemotherapy plus Single-Agent Intrathecal Chemotherapy followed by 2-Drug Combination Systemic Chemotherapy. DM/VCR/MTX/MP; plus IT ARA-C followed by VP-16/CTX/Mesna. ROUTINE MAINTENANCE: 4-Drug Combination Systemic Chemotherapy plus Single-Agent Intrathecal Chemotherapy. VCR/MTX/MP/PRED; plus IT MTX. TRANSPLANTATION: 2-Drug Combination Myeloablative Chemotherapy followed by Radiotherapy followed by Hematopoietic Rescue plus GVHD Prophylaxis. ARA-C/CTX; followed by TBI using a linear accelerator or Co60 equipment; followed by AlBM; plus MePRDL; CYSP.

PROJECTED ACCRUAL: 100 patients per year will be entered over approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed acute lymphoblastic leukemia (ALL) in infants under 12 months of age at diagnosis Adequate bone marrow and/or peripheral blood specimens with blasts available No prior treatment for ALL except emergency therapy for the following: Blast cell crisis Superior vena cava syndrome Renal failure due to leukemic infiltration of the kidneys

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1996-07; Primary Completion 2000-08 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Dinndorf, MD, Study Chair — Children's National Research Institute
Locations (33):
- United States (30):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Dreyer ZE, Dinndorf PA, Camitta B, Sather H, La MK, Devidas M, Hilden JM, Heerema NA, Sanders JE, McGlennen R, Willman CL, Carroll AJ, Behm F, Smith FO, Woods WG, Godder K, Reaman GH. Analysis of the role of hematopoietic stem-cell transplantation in infants with acute lymphoblastic leukemia in first remission and MLL gene rearrangements: a report from the Children's Oncology Group. J Clin Oncol. 2011 Jan 10;29(2):214-22. doi: 10.1200/JCO.2009.26.8938. Epub 2010 Dec 6. PMID 21135279
- [Background] Nguyen K, Devidas M, Cheng SC, La M, Raetz EA, Carroll WL, Winick NJ, Hunger SP, Gaynon PS, Loh ML; Children's Oncology Group. Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia. 2008 Dec;22(12):2142-50. doi: 10.1038/leu.2008.251. Epub 2008 Sep 25. PMID 18818707
- [Result] Salzer W, Dinndorf P, Dreyer Z, Hilden J, Reaman GH. Analysis of infectious complications in infants with acute lymphoblastic leukemia treated on the Children's Cancer Group Protocol 1953: a report from the Children's Oncology Group. J Pediatr Hematol Oncol. 2009 Jun;31(6):398-405. doi: 10.1097/MPH.0b013e3181a6dec0. PMID 19648788
- [Result] Robinson BW, Cao K, Hilden JM, et al.: Age is the strongest determinant of leukemia blast cell gene expression in MLL-rearranged infant ALL and MLL-AF4 directs a distinct gene expression profile related to CNS disease. [Abstract] Blood 112 (11): A-1200, 2008.
- [Result] Hilden JM, Dinndorf PA, Meerbaum SO, Sather H, Villaluna D, Heerema NA, McGlennen R, Smith FO, Woods WG, Salzer WL, Johnstone HS, Dreyer Z, Reaman GH; Children's Oncology Group. Analysis of prognostic factors of acute lymphoblastic leukemia in infants: report on CCG 1953 from the Children's Oncology Group. Blood. 2006 Jul 15;108(2):441-51. doi: 10.1182/blood-2005-07-3011. Epub 2006 Mar 23. PMID 16556894